CLINICAL TRIAL: NCT03359733
Title: An Open-Label, Phase 1, Two-Way, Crossover Study of the Effect of Food on the Pharmacokinetics of TAK-659 in Patients With Advanced Solid Tumor and/or Lymphoma Malignancies
Brief Title: A Study to Evaluate the Effect of Food on the Pharmacokinetics (PK) of TAK-659 in Participants With Advanced Solid Tumor
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision: no safety or efficacy concerns
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C34009; U1111-1201-1081 (Registry Identifier: WHO)
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Lymphoma, Malignant; Advanced Solid Neoplasms
Keywords: Drug therapy
MeSH Terms: conditions — Lymphoma | interventions — TAK-659

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAK-659 100 mg Fasted + TAK-659 100 mg Fed (Experimental): TAK-659 100 milligram (mg), tablet, orally under fasted state, once on Day 1, followed by TAK-659 100 mg, tablet, orally under fed state, once on Day 8 of a 15-day food effect treatment period.
  Interventions: Drug: TAK-659
- TAK-659 100 mg Fed + TAK-659 100 mg Fasted (Experimental): TAK-659 100 mg, tablet, orally under fed state, once on Day 1, followed by TAK-659 100 mg, tablet, orally under fasted state, once on Day 8 of a 15-day food effect treatment period.
  Interventions: Drug: TAK-659

INTERVENTIONS:
Drug: TAK-659 — TAK-659 tablet.

SUMMARY:
The purpose of this study is to characterize the effect of food on the single-dose PK of TAK-659 in participants with advanced solid tumors and/or lymphomas.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-659. TAK-659 is being tested in participants with advanced solid tumors and/or lymphomas in order to determine the effect of food on the PK of single oral dose of TAK-659 tablet formulation. The study will enroll approximately 20 participants. Participants will be randomly and equally assigned (by chance, like flipping a coin) to 1 of the 2 treatment sequences following as:

* TAK-659 100 mg Fasted + TAK-659 100 mg Fed
* TAK-659 100 mg Fed + TAK-659 100 mg Fasted

All participants will be asked to take single oral dose of TAK-659 tablet on Day 1 and Day 8 of a 15-day food effect treatment period. Upon completion of the food effect treatment period, participants can continue in the optional post food effect treatment period to receive TAK-659 100 mg, once daily in a 28-day treatment cycle until disease progression, unacceptable toxicity, or the start of another anticancer therapy upon request by the investigator and agreement by the project clinician.

This single or multi-center trial will be conducted in the United States. The overall time to participate in this study is up to 58 weeks. Participants will visit the clinic on Day -1 and remain confined until Day 15 of food effect treatment period. Participants will make a visit to the clinic after 28 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a histologically or cytologically confirmed metastatic and/or advanced solid tumor and/or lymphoma for which standard curative or life-prolonging treatment does not exist, or is no longer effective or tolerable.
2. Has an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
3. Has a life expectancy of at least 3 months.
4. Suitable venous access for the study-required blood sampling (that is, PK).
5. Must have adequate organ function, including the following:

   * Adequate bone marrow reserve: absolute neutrophil count (ANC) greater than or equal to (>=) 1000 per cubic millimeter (/mm^3), platelet count >=75,000/ mm^3 (>=50,000 per micro liter (/mcL) for participants with bone marrow involvement), and hemoglobin >=8 gram per deciliter (g/dL) (red blood cell [RBC] transfusion allowed >=14 days before assessment).
   * Hepatic: total bilirubin less than or equal to (<=) 1.5*the upper limit of the normal range (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=2.5*ULN.
   * Renal: serum creatinine <=1.5*ULN or creatinine clearance >=60 milliliter per minute (mL/min) as estimated by the Cockcroft-Gault equation or based on urine collection (12 or 24 hours).

Exclusion Criteria:

1. Central nervous system (CNS) lymphoma; active brain or leptomeningeal metastases, as indicated by positive cytology from lumbar puncture or computed tomography (CT) scan/magnetic resonance imaging (MRI).
2. History of drug-induced pneumonitis requiring treatment with steroids; history of idiopathic pulmonary fibrosis, organizing pneumonia, or evidence of active pneumonitis on screening chest CT scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted.
3. Systemic anticancer treatment (including investigational agents) less than 3 weeks before the first dose of study treatment (<=4 weeks for antibody-based therapy including unconjugated antibody, antibody-drug conjugate, and bi-specific T-cell engager agent; <=8 weeks for cell-based therapy or anti-tumor vaccine).
4. Radiotherapy less than 3 weeks before the first dose of study treatment.
5. Use or consumption of any of the following substances:

   * Medications or supplements that are known to be inhibitors of P-glycoprotein (P-gp) and/or strong reversible inhibitors of cytochrome P450 (CYP) 3A within 5*the inhibitor half-life (if a reasonable half-life estimate is known), or within 7 days (if a reasonable half-life estimate is unknown), before the first dose of study drug.
   * Medications or supplements that are known to be strong CYP3A mechanism-based inhibitors or strong CYP3A inducers and/or P-gp inducers within 7 days or within 5 times the inhibitor or inducer half-life (whichever is longer) before the first dose of study drug. In general, the use of these agents is not permitted during the study except in cases in which an AE must be managed during interruption of study drug dosing.
   * Food or beverages containing grapefruit within 5 days before the first dose of study drug. Note that food and beverages containing grapefruit are not permitted during the study.
6. Major surgery within 14 days before the first dose of study drug and not recovered fully from any complications from surgery.
7. Active secondary malignancy that requires treatment. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection and are considered disease-free at the time of study entry.
8. Lactose-intolerance or are unwilling/unable to consume the protocol-specified standardized high-fat, high-calorie breakfast.
9. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of TAK-659, including difficulty swallowing tablets or diarrhea greater than (>) Grade 1 despite supportive therapy.
10. Treatment with high-dose corticosteroids for anticancer purposes within 14 days before the first dose of TAK-659; daily dose equivalent to 10 mg oral prednisone or less is permitted. Corticosteroids for topical use or in nasal spray or inhalers are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-28 (Estimated); Primary Completion 2019-01-14 (Estimated); Study Completion 2019-08-20 (Estimated)

PRIMARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for TAK-659 | Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-659 | Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-659 | Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Cmax: Maximum Observed Plasma Concentration for TAK-659 | Day 8 pre-dose and at multiple time points (up to 168 hours) post-dose
AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-659 | Day 8 pre-dose and at multiple time points (up to 168 hours) post-dose
AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-659 | Day 8 pre-dose and at multiple time points (up to 168 hours) post-dose

SECONDARY OUTCOMES:
Percentage of Participants Reporting one or More Treatment-emergent Adverse Events (TEAEs) | Baseline up to 28 days after the last dose of study drug (up to 58 weeks)
Percentage of Participants With Grade 3 or Above Adverse Event (AE) | Baseline up to 28 days after the last dose of study drug (up to 58 weeks)
  AE Grades will be evaluated as per National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE), version 4.03. Grade 1 scaled as Mild; Grade 2 scaled as Moderate; Grade 3 scaled as severe or medically significant but not immediately life-threatening; Grade 4 scaled as life-threatening consequences; and Grade 5 scaled as death related to AE.
Percentage of Participants With Drug-related AEs | Baseline up to 28 days after the last dose of study drug (up to 58 weeks)
Percentage of Participants With Drug-related Grade 3 or Above AEs | Baseline up to 28 days after the last dose of study drug (up to 58 weeks)
  AE Grades will be evaluated as per NCI CTCAE, version 4.03. Grade 1 scaled as Mild; Grade 2 scaled as Moderate; Grade 3 scaled as severe or medically significant but not immediately life-threatening; Grade 4 scaled as life-threatening consequences; and Grade 5 scaled as death related to AE.
Percentage of Participants who Experience at Least 1 Serious Adverse Event (SAE) | Baseline up to 28 days after the last dose of study drug (up to 58 weeks)
Percentage of Participants who Discontinue due to an AE | Baseline up to 28 days after the last dose of study drug (up to 58 weeks)
Percentage of Participants who Meet the Takeda Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post Dose | Baseline up to 28 days after the last dose of study drug (up to 58 weeks)
Percentage of Participants who Meet the Takeda Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post Dose | Baseline up to 28 days after the last dose of study drug (up to 58 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Yale Cancer Center, New Haven, Connecticut
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Montefiore Medical Center, The Bronx, New York